CLINICAL TRIAL: NCT03793868
Title: Perampanel Single Ascending Dose Transcranial Magnetic Stimulation Biomarker Study in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bjorn E. Oskarsson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-002396
Record Dates: First submitted 2018-12-28; First posted 2019-01-04 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — perampanel

STUDY DESIGN:
Intervention Model Description: This is a pilot study for the assessment of transcranial magnetic stimulation as a biomarker for ALS and to obtain information to guide a dose selection for future biomarker driven Phase 2 studies of Perampanel in ALS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose (Experimental): Perampanel 4mg PO x1
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): Receiving placebo
  Interventions: Other: Placebo
- High dose (Experimental): Perampanel 8 mg PO x1
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Oral tablet
  Other Names: Fycompa
  Arms: High dose; Low dose
Other: Placebo — Placebo (not drug)
  Arms: Placebo

SUMMARY:
To evaluate if transcranial magnetic stimulation can be used as a biomarker in Amyotrophic Lateral sclerosis (ALS).

DETAILED DESCRIPTION:
To measure the effect on motor threshold (MT) by transcranial magnetic stimulation (TMS) after a single dose of perampanel at two dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. A probable laboratory supported, probable or definitive ALS diagnosis by revised El Escorial criteria.
2. Sporadic or familial ALS.
3. Ages of 18-70.
4. Agree to use reliable contraception
5. Randomization will occur after a baseline MT has been established; any subject in whom a MT cannot be established will be excluded.
6. Caregiver willing to report adverse behavioral events. -

Exclusion Criteria:

1. History of epilepsy.
2. Significant laboratory abnormality (AST or alanine aminotransferase >3x upper limit of normal, or glomerular filtration rate <60)
3. History of aggressive behavior.
4. Subject unwilling to abstain from alcohol for 2 weeks after each dosing.
5. History of drug abuse in the last 5 years
6. Other severe medical conditions, including psychiatric conditions, which would cause an increased risk in the opinion of the investigator, including but not limited to renal failure and liver failure.
7. Skull defect or other physical contraindication for TMS
8. Pacemaker or implanted defibrillator
9. Inability to take study capsule by mouth

Females only: Subject is pregnant [as confirmed by a positive serum human chorionic gonadotropin (hCG) test for females of reproductive potential (FRP) only], subject is breastfeeding, or subject is of reproductive potential and does not agree to follow use of reliable contraception.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Motor threshold (MT) | at 4 hours post dose
  Transcranial Magnetic stimulation motor threshold change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn E Oskarsson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Oskarsson B, Mauricio EA, Shah JS, Li Z, Rogawski MA. Cortical excitability threshold can be increased by the AMPA blocker Perampanel in amyotrophic lateral sclerosis. Muscle Nerve. 2021 Aug;64(2):215-219. doi: 10.1002/mus.27328. Epub 2021 May 27. PMID 34008857
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials